CLINICAL TRIAL: NCT04992065
Title: Dose Response and Safety of an Oral PCSK9i, NNC0385-0434, in Patients With Established Atherosclerotic Cardiovascular Disease (ASCVD) or ASCVD Risk on Maximally Tolerated Statin Dose and Other Lipid-lowering Therapy Requiring Further LDL-C Reduction
Brief Title: A Research Study Looking at How NNC0385-0434 Tablets Work to Lower Blood Cholesterol in People With Heart Disease or a High Risk of Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN6435-4697; U1111-1252-3392 (Other: World Health Organization (WHO)); 2020-002630-32 (EudraCT Number); 151409 (Other: IND Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The trial will be double-blinded within dose level of oral NNC0385-0434 and size-matched placebo arm. The subcutaneous (s.c.) evolocumab arm will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Oral NNC0385-0434 15 mg once-daily (OD) (Experimental): 15 mg NNC0385-0434 co-formulated with 500 mg Salcaprozate sodium (SNAC) tablet once daily
  Interventions: Drug: NNC0385-0434 A 15 mg
- Oral placebo (NNC0385-0434 15 mg) (Placebo Comparator): 15 MG placebo administered as tablets (without SNAC) once daily
  Interventions: Other: Placebo I A (for NNC0385-0434 A 15 mg)
- Oral NNC0385-0434 40 mg OD (Experimental): 40 mg study drug co-formulated with 500 mg SNAC tablet once daily
  Interventions: Drug: NNC0385-0434 A 40 mg
- Oral placebo (NNC0385-0434 40 mg) (Placebo Comparator): placebo administered as tablets (without SNAC) once daily
  Interventions: Other: Placebo I A (for NNC0385-0434 A 40 mg)
- Oral NNC0385-0434 100 mg (Experimental): 100 mg NNC0385-0434 co-formulated with 500 mg SNAC tablet once daily (51 participants)
  Interventions: Drug: NNC0385-0434 A 100 mg
- Oral placebo (NNC0385-0434 100 mg) (Placebo Comparator): placebo administered as tablets (without SNAC) once daily
  Interventions: Other: Placebo II A (for NNC0385-0434 A 100 mg)
- Subcutaneous evolocumab 140 mg Q2W (Active Comparator): 140 mg evolocumab Subcutaneous (s.c.) injections every 2 weeks (51 participants). The s.c. evolocumab arm is open-label to limit unnecessary injections
  Interventions: Drug: Evolocumab 140 mg/mL, Repatha®

INTERVENTIONS:
Drug: NNC0385-0434 A 15 mg — 15 mg administered as one oral tablet once daily in the morning in a fasting state. The tablet should be taken at least 30 min before the first food, beverage or other oral medications of the day. The tablet can be taken with up to half a glass of water (approximately 120 mL/ 4 fluid ounces).
  Arms: Oral NNC0385-0434 15 mg once-daily (OD)
Drug: NNC0385-0434 A 40 mg — 40 mg administered as one oral tablet once daily in the morning in a fasting state. The tablet should be taken at least 30 min before the first food, beverage or other oral medications of the day. The tablet can be taken with up to half a glass of water (approximately 120 mL/ 4 fluid ounces).
  Arms: Oral NNC0385-0434 40 mg OD
Other: Placebo I A (for NNC0385-0434 A 15 mg) — Placebo administered as 1 tablet once daily in the morning in a fasting state. The tablet should be taken at least 30 min before the first food, beverage or other oral medications of the day. The tablet can be taken with up to half a glass of water (approximately 120 mL/ 4 fluid ounces). placebo tablets are sized match to the active arm within dose level
  Arms: Oral placebo (NNC0385-0434 15 mg)
Drug: NNC0385-0434 A 100 mg — 100 mg administered as one oral tablet once daily in the morning in a fasting state.
  The tablet should be taken at least 30 min before the first food, beverage or other oral medications of the day.
  The tablet can be taken with up to half a glass of water (approximately 120 mL/ 4 fluid ounces).
  Arms: Oral NNC0385-0434 100 mg
Other: Placebo I A (for NNC0385-0434 A 40 mg) — Placebo administered as one tablet once daily in the morning in a fasting state.
  The tablet should be taken at least 30 min before the first food, beverage or other oral medications of the day.
  The tablet can be taken with up to half a glass of water (approximately 120 mL/ 4 fluid ounces).
  placebo tablets are sized match to the active arm within dose level
  Arms: Oral placebo (NNC0385-0434 40 mg)
Other: Placebo II A (for NNC0385-0434 A 100 mg) — Placebo administered as one tablet once daily in the morning in a fasting state.
  The tablet should be taken at least 30 min before the first food, beverage or other oral medications of the day.
  The tablet can be taken with up to half a glass of water (approximately 120 mL/ 4 fluid ounces).
  placebo tablets are sized match to the active arm within dose level
  Arms: Oral placebo (NNC0385-0434 100 mg)
Drug: Evolocumab 140 mg/mL, Repatha® — Every 2 weeks subcutaneous (s.c.) injection of 140 mg into areas of the abdomen, thigh, or upper arm that are not tender, bruised, red, or indurated. Administered using a pre-filled SureClick® autoinjector (single-use).
  Dose volume: 1 mL
  Arms: Subcutaneous evolocumab 140 mg Q2W

SUMMARY:
This study looks at how well a new medicine, NNC0385-0434, works to lower blood cholesterol levels. Participants will either get NNC0385-0434 as a tablet (a potential new medicine), or placebo as a tablet (a dummy medicine that looks like NNC0385-0434 but has no effect on the body), or evolocumab as an injection (a medicine that doctors can already prescribe).

Which treatment participants get is decided by chance. If participants get NNC0385-0434 or placebo participants will need to take 1 tablet every morning. If participants get evolocumab participants will need to take 1 injection every 2 weeks.

The study will last for about 22 weeks. About 255 people will participate in the study. Participants will have 9 visits to the clinic and 2 phone calls with the study doctor. Some people will be invited to participate in a sub-study and will have 4 extra visits (13 visits in total). Participants will have blood samples taken at all visits to the clinic (except visit 0). At 4 clinic visits, participants will have an electrocardiogram (ECG). This is a test to check your heart.

Women can only take part in the study if they are not able to become pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential.
* Established atherosclerotic cardiovascular disease (ASCVD) (criteria a) or ASCVD risk (criteria b):

  1. Age 40 years or older at the time of signing informed consent and history of ASCVD
  2. Age above 50 years at the time of signing informed consent and with ASCVD risk
* Serum LDL-C above or equal to 1.8 mmol/L (above or equal to 70 mg/dL) as measured by the central laboratory at screening.
* Japanese participants: Serum LDL-C above or equal to 2.6 mmol/L (above or equal to 100 mg/dL) for participants of 40 years of age or older and with a history of coronary heart disease, and serum LDL-C above or equal to 3.1 mmol/L (above or equal to 120 mg/dL) for all other Japanese participants
* Participants must be on maximally tolerated dose of statins.
* Participants not receiving statin must have documented evidence of intolerance to all doses of at least two different statins.

Exclusion Criteria:

* Treatment with PCSK9i therapy (alirocumab or evolocumab within 90 days prior to screening) or PCSK9 siRNA therapy (inclisiran within 12 months prior to screening).
* Fasting triglyceride above 4.52 mmol/L (above 400 mg/dL) as measured by the central laboratory at screening.
* Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Renal impairment with eGFR less than 30 ml/min/1.73 m2 as measured by the central laboratory at screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (44):
- United States (13):
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Excel Med Ctr Clinical Trials, Boca Raton, Florida
  - Integrative Research Associates, Inc, Fort Lauderdale, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Northwest Heart Clin. Res., Arlington Heights, Illinois
  - Louisiana Heart Center, Covington, Louisiana
  - Louisiana Heart Center_Slidell, Slidell, Louisiana
  - VA NEB - Western IA Health Stm, Omaha, Nebraska
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Albany Medical College - Endo, Albany, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Thyroid, Endocrinology, and Diabetes, PA, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
- Belgium (5):
  - Algemeen Stedelijk Ziekenhuis - Aalst - Interventional Cardiology, Aalst
  - AZ Sint-Jan - Campus Brugge, Bruges
  - Ziekenhuis Oost-Limburg AV - Cardiology, Genk
  - Hôpital de Jolimont_Haine-Saint-Paul_0, Haine-Saint-Paul
  - Jessa Ziekenhuis - Hasselt - Cardiology, Hasselt
- Germany (4):
  - MVZ CCB Frankfurt Und Main-Taunus GbR, Frankfurt
  - Medical Center - University Of Freiburg, Freiburg im Breisgau
  - Deutsches Herzzentrum München - Klinik für Herz- und Kreislauferkrankungen, München
  - Jacob, Villingen-Schwenningen, Villingen-Schwenningen
- Greece (6):
  - "Sotiria" Thoracic Diseases Hospital of Athens, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - U.G.H of Athens "Attikon", Chaidari, Athens
  - General Hospital of Chios "Skilitsio", Chios
- Japan (4):
  - Sanai Hospital, Saitama-shi, Saitama
  - Shinden Higashi Clinic, Sendai-shi, Miyagi
  - Soka Sugiura Internal Medicine Clinic, Soka-shi, Saitama
  - Minamino Cardiovascular Hospital, Tokyo
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Deventer Ziekenhuis, Deventer
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Haarlem
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - D & A Research B.V., Sneek
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Regionalny Osrodek Kardiologii, Lubin
  - Lubelskie Centrum Diagnostyczne Tomasz Blicharski, Świdnik
  - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
  - Szpital Grochowski im. dr med. Rafała Masztaka Sp. z o.o., Warsaw
  - Narodowy Instytut Kardiologii Stefana kardynała Wyszynskiego, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Koren MJ, Descamps O, Hata Y, Hengeveld EM, Hovingh GK, Ikonomidis I, Radu Juul Jensen MD, Langbakke IH, Martens FMAC, Sondergaard AL, Witkowski A, Koenig W. PCSK9 inhibition with orally administered NNC0385-0434 in hypercholesterolaemia: a randomised, double-blind, placebo-controlled and active-controlled phase 2 trial. Lancet Diabetes Endocrinol. 2024 Mar;12(3):174-183. doi: 10.1016/S2213-8587(23)00325-X. Epub 2024 Feb 1. PMID 38310920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 7 countries as follows (number of sites that screened participants/ number of sites that randomized participants): Belgium (5/5), Germany (4/4), Greece (6/6), Japan (4/4), Netherlands (6/6), Poland (5/5)and United States (12/12).
Groups:
- NNC0385-0434 15 mg: Participants received 15 milligrams (mg) NNC0385-0434 (co-formulated with 500 mg salcaprozate sodium [SNAC]) tablet orally once daily for 12 weeks.
- NNC0385-0434 40 mg: Participants received 40 mg NNC0385-0434 (co-formulated with 500 mg SNAC) tablet orally once daily for 12 weeks.
- NNC0385-0434 100 mg: Participants received 100 mg NNC0385-0434 (co-formulated with 500 mg SNAC) tablet orally once daily for 12 weeks.
- Placebo: Participants received placebo matched to NNC0385-0434 (without SNAC) tablet orally once daily for 12 weeks.
- Evolocumab 140 mg: Participants received 140 mg evolocumab subcutaneously (s.c.) every 2 weeks for 12 weeks.
Period: Overall Study
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Started | 53 | 53 | 53 | 54 | 54
Treated | 53 | 53 | 53 | 54 | 54
Full Analysis Set | 53 | 53 | 53 | 54 | 54
Safety Analysis Set | 53 | 53 | 53 | 54 | 54
Completed | 53 | 53 | 53 | 54 | 54
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg | Total
Number analyzed (Participants) | 53 | 53 | 53 | 54 | 54 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (9.3) | 64.6 (8.6) | 65.2 (9.2) | 63.1 (8.6) | 64.5 (9.6) | 64.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 14 | 17 | 17 | 82
  Male | 36 | 36 | 39 | 37 | 37 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 53 | 53 | 53 | 52 | 53 | 264
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 7 | 5 | 5 | 7 | 6 | 30
  Race: Black or African American | 0 | 4 | 4 | 1 | 2 | 11
  Race: White | 46 | 44 | 44 | 46 | 46 | 226
  Race: Other | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Low-density Lipoprotein (LDL)-Cholesterol
Description: Percentage change in LDL-cholesterol (LDL-C) (measured in milligrams per deciliter [mg/dL]) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period. The in-trial period is defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
Time Frame: Baseline (week 0), week 12
Population: FAS included all randomized participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change of LDL cholesterol
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 51 | 52 | 49 | 52 | 49
Percentage change of LDL cholesterol | -27 (19) | -41 (37) | -55 (20) | 6 (41) | -59 (22)
Statistical Analysis 1: Comparison: NNC0385-0434 15 mg vs Placebo; LDL-C percentage change at week 12 from baseline responses were analysed using an analysis of covariance model with randomised treatment and strata as factors and baseline LDL-C as covariate; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -31.95, 95% CI 2-sided [-43.02 to -20.87]
Statistical Analysis 2: Comparison: NNC0385-0434 40 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -44.91, 95% CI 2-sided [-56.04 to -33.79]
Statistical Analysis 3: Comparison: NNC0385-0434 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -61.83, 95% CI 2-sided [-72.94 to -50.72]
Statistical Analysis 4: Comparison: NNC0385-0434 15 mg vs Evolocumab 140 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Treatment difference = 33.32, 95% CI 2-sided [22.16 to 44.47]
Statistical Analysis 5: Comparison: NNC0385-0434 40 mg vs Evolocumab 140 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Treatment difference = 20.35, 95% CI 2-sided [9.21 to 31.48]
Statistical Analysis 6: Comparison: NNC0385-0434 100 mg vs Evolocumab 140 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Treatment difference = 3.43, 95% CI 2-sided [-7.81 to 14.68]

2. Secondary Outcome: Percentage Change in Total Cholesterol
Description: Percentage change in total cholesterol (measured in millimoles per iliter [mmol/L]) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of total cholesterol
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 52 | 52 | 50 | 53 | 52
Percentage change of total cholesterol | -14 (13) | -25 (27) | -33 (11) | 4 (23) | -38 (14)

3. Secondary Outcome: Percentage Change in High Density Lipoprotein (HDL)-Cholesterol
Description: Percentage change in HDL-cholesterol (measured in mg/dL) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of HDL cholesterol
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 52 | 52 | 47 | 53 | 51
Percentage change of HDL cholesterol | 4 (13) | 5 (16) | 7 (16) | 1 (14) | 5 (14)

4. Secondary Outcome: Percentage Change in Very Low Density Lipoprotein (VLDL)-Cholesterol
Description: Percentage change in VLDL-cholesterol (measured in mmol/L) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of VLDL cholesterol
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 52 | 52 | 50 | 53 | 52
Percentage change of VLDL cholesterol | 5 (27) | -7 (33) | -15 (26) | 3 (41) | -16 (24)

5. Secondary Outcome: Percentage Change in Triglycerides
Description: Percentage change in triglycerides (measured in mg/dL) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of triglycerides
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 52 | 52 | 50 | 53 | 52
Percentage change of triglycerides | 5 (27) | -7 (31) | -16 (27) | 2 (41) | -16 (23)

6. Secondary Outcome: Percentage Change in Total Apolipoprotein B (Apo B)
Description: Percentage change in Apo B (measured in mg/dL) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of Apo B
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 51 | 52 | 49 | 53 | 53
Percentage change of Apo B | -20 (15) | -34 (28) | -48 (12) | 6 (31) | -52 (17)

7. Secondary Outcome: Percentage Change in Total Apolipoprotein CIII (Apo CIII)
Description: Percentage change in Apo CIII (measured in mg/dL) at week 12 is presented. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of Apo CIII
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 50 | 52 | 48 | 51 | 52
Percentage change of Apo CIII | -0 (20) | -7 (24) | -16 (15) | 2 (23) | -15 (21)

8. Secondary Outcome: Change in Total Lipoprotein(a) (Lp[a]): Ratio to Baseline
Description: Change in total Lp(a) (measured in mg/dL) at week 12 is presented as ratio to baseline. Data is reported for the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: Baseline (week 0), week 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Lipoprotein (a)
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 52 | 52 | 50 | 53 | 53
Ratio of Lipoprotein (a) | 0.79 (34.2) | 0.70 (37.6) | 0.66 (40.0) | 0.99 (31.5) | 0.59 (43.4)

9. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse events (AE) is any untoward medical occurrence in a clinical trial participant that is temporally associated with the use of an investigational medicinal product (IMP), whether or not considered related to the IMP. All presented AEs are TEAEs. TEAEs was the number of AEs recorded during the on-treatment period. The on-treatment period is the time period where participants were considered exposed to trial product. The observation period starts at the date of first dose of trial product and ends at the first date of any of the following: The follow-up visit or the last date on randomised treatment regimen + 58 days or the end-date for the 'in-trial' observation period.
Time Frame: From baseline (week 0) to 138 days
Population: Safety analysis set (SAS) included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Measure: Number; unit: Events
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
Number analyzed (Participants) | 53 | 53 | 53 | 54 | 54
Events | 82 | 60 | 65 | 56 | 81

ADVERSE EVENTS:
Time Frame: Up to 138 Days
Description: All presented AEs are TEAEs. TEAEs: AEs recorded during on-treatment period. SAS included all participants randomly assigned to trial treatment who took at least 1 dose of trial product. On-treatment period: time period where participants were exposed to trial product. Observation period starts at date of first dose of trial product and ends at first date of any of following: follow-up visit or last date on randomised treatment regimen + 58 days or end-date for 'in-trial' observation period.
Arm/Group | NNC0385-0434 15 mg | NNC0385-0434 40 mg | NNC0385-0434 100 mg | Placebo | Evolocumab 140 mg
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53 | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 1/53 | 3/53 | 1/53 | 5/54 | 3/54
Other Adverse Events (participants affected / at risk) | 16/53 | 14/53 | 19/53 | 14/54 | 17/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC0385-0434 15 mg (N=53) | NNC0385-0434 40 mg (N=53) | NNC0385-0434 100 mg (N=53) | Placebo (N=54) | Evolocumab 140 mg (N=54)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC0385-0434 15 mg (N=53) | NNC0385-0434 40 mg (N=53) | NNC0385-0434 100 mg (N=53) | Placebo (N=54) | Evolocumab 140 mg (N=54)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 8 (8) | 8 (8) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 2 (5) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT04992065/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT04992065/SAP_001.pdf